CLINICAL TRIAL: NCT06824311
Title: Clinical Characteristics and Outcome of Patients with Hemorrhagic Stroke Admitted in Neurology Department in a Tertiary Hospital
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Sumit Shahi, Resident, Department of Neurology, Principal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 437 (6-11) E2
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Hemorrhage, Intracranial; Outcome Measure
Keywords: hemorrhagic stroke; spontaneous intracerebral hemorrhage; mRS scale; functional outcome after stroke
MeSH Terms: conditions — Intracranial Hemorrhages; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main aim of this study is to know about the clinical profile of patients who are diagnosed as hemorrhagic stroke as well as the factors that affect good and bad outcomes of those patients after 3 months. Patients will be required to follow up in medical OPD of the same institution after 3 months.

DETAILED DESCRIPTION:
This was a prospective observational study conducted on 197 patients of ≥ 18 years of age admitted with the diagnosis of hemorrhagic stroke in Tribhuvan University Teaching Hospital, a tertiary hospital in Nepal from April 1 2023 to March 31, 2024. Patients who do not give consent or with post-traumatic hemorrhages, hemorrhagic transformation of an ischemic stroke, or any intracranial hemorrhages other than primary intracranial hemorrhages were excluded from the study. The study protocol and design were reviewed and approved by the Institutional Review Committee of Tribhuvan University Teaching Hospital [Ref. 437 (6-11) E2]. Data was collected in a structured proforma.

The primary outcome of this study was to assess the functional outcome of the patients at 3 months of follow-up. The modified Rankin scale (mRS) was assessed in an outpatient setting during the follow-up. If patients did not attend the 3-month follow-up, mRS was assessed by telephone conversation. Clinical outcome was dichotomously categorized as good outcome if mRS was 0-2 and bad outcome if mRS was ≥ 3.

Analysis for categorical data was done by Chi-squared test, Fisher's exact test. Analysis for continuous data was done using either parametric tests like the t-test, or non-parametric tests like the Mann-Whitney U test depending on the distribution of data. Predictors of clinical outcomes were analyzed using multivariate logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed case of hemorrhagic stroke

Exclusion Criteria:

* Does not give consent
* Post-traumatic hemorrhages, hemorrhagic transformation of an ischemic stroke, or any intracranial hemorrhages other than primary intracranial hemorrhages were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in neurology department of Tribhuvan University Teaching Hospital with diagnosis of hemorrhagic stroke
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale at 3 months | From the diagnosis of hemorrhagic stroke to 3 months of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Maharajgunj, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaik MM, Loo KW, Gan SH. Burden of stroke in Nepal. Int J Stroke. 2012 Aug;7(6):517-20. doi: 10.1111/j.1747-4949.2012.00799.x. Epub 2012 Jun 13. PMID 22691158
- [Background] Feigin VL, Brainin M, Norrving B, Martins S, Sacco RL, Hacke W, Fisher M, Pandian J, Lindsay P. World Stroke Organization (WSO): Global Stroke Fact Sheet 2022. Int J Stroke. 2022 Jan;17(1):18-29. doi: 10.1177/17474930211065917. PMID 34986727
- [Background] Katan M, Luft A. Global Burden of Stroke. Semin Neurol. 2018 Apr;38(2):208-211. doi: 10.1055/s-0038-1649503. Epub 2018 May 23. PMID 29791947